CLINICAL TRIAL: NCT01064700
Title: Bright Light: A Novel Treatment for Anxiety
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of South Carolina (Other)
Collaborators: Liteboook Company (Unknown)
Responsible Party: Principal Investigator, Shawn Youngstedt, Assistant Professor, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HSA-3469
Record Dates: First submitted 2010-02-04; First posted 2010-02-08 (Estimated); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Anxiety; Depression; Sleep
Keywords: Anxiety; Phototherapy; Psychic Anxiety
MeSH Terms: conditions — Anxiety Disorders; Depression | interventions — Phototherapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Baseline (No Intervention): 1 week period, in which subjects followed usual schedule, though they were asked to maintain a fairly stable sleep schedule. The baseline period was used for comparison with the experimental intervention.
- Experimental Intervention (Experimental): Randomized exposure to the 4-week experimental treatments.
  Interventions: Device: Litebook Bright Light Box; Device: Litebook inactivated negation ion generator (the placebo)

INTERVENTIONS:
Device: Litebook Bright Light Box — Four weeks of daily exposure to bright light (3,000 lux) for 45 min/day, beginning within 60 min of arising.
  Other Names: Phototherapy
  Arms: Experimental Intervention
Device: Litebook inactivated negation ion generator (the placebo) — Four weeks of daily exposure to inactivated negative ion generator for 45 min/day, beginning within 60 min of arising
  Other Names: Placebo
  Arms: Experimental Intervention

SUMMARY:
The primary aim of this research was to examine the influence of bright light on anxiety in high-anxious young adults. In an acute exposure study, participants were randomly assigned to 45 min of either (1) bright light (3,000 lux) or (2) a placebo inactivated negative ion generator. Treatments were initiated ≤1 hr after awakening. At 10 min before and 30 min after the treatments, state anxiety, mood, and blood pressure were assessed.

Following the acute exposure study, participants performed a 5-week study. Following a a 1-week baseline, participants were randomly assigned to four weeks of daily exposure to either (1) bright light (45 min/day; 3,000 lux) or (2) placebo inactivated negative ion generator, which were initiated ≤1 hr after awakening. Before and after the experiment, clinical ratings were conducted with the Hamilton Anxiety Scale, the Hamilton Depression Scale, and the Clinical Global Impressions scale (CGI). Following baseline, and following each week of treatment, blood pressure, as well as questionnaires for state anxiety, depression, mood, sleep, and side effects were assessed.

ELIGIBILITY:
Inclusion Criteria:

* Having a level of trait anxiety [Spielberger State-Trait Anxiety Inventory (Form Y1)]{23642} that was ≥ the 75th percentile for their age (i.e., ≥ 46 and ≥ 44 for women and men, respectively)

Exclusion Criteria:

* Current treatment for anxiety or depression;
* History of bipolar disorder, mania, or psychotic disorders;
* History of winter depression, which might bias towards positive response to light;
* Hypertension;
* Ophthalmic abnormalities; and
* Usual exposure to high levels of light such that the intervention would add little to usual exposure.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2006-10; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Spielberger State Anxiety Inventory | 5 weeks
  state anxiety questionnaire
Hamilton Anxiety | 5 weeks
  Hamilton Anxiety Questionnaire

SECONDARY OUTCOMES:
Beck Depression Inventory | 5 weeks
  self-report depression questionnaire
Pittsburgh Sleep Quality Inventory | 5 weeks
  PSQI, a common sleep quality questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Shawn D Youngstedt, Principal Investigator — University of Southern California
Locations (1):
- Chronobiology Lab, University of South Carolina, Columbia, South Carolina, United States

REFERENCES:
- [Derived] Youngstedt SD, Kline CE, Ginsberg JP, Zielinski MR, Hardin JW. Bright light treatment for high-anxious young adults: a randomized controlled pilot study. Depress Anxiety. 2011 Apr;28(4):324-32. doi: 10.1002/da.20784. Epub 2011 Jan 19. PMID 21254315